CLINICAL TRIAL: NCT04562519
Title: Hyposalivation Response to TENS in HD Patients
Brief Title: Salivary Flow Rate Response to Electrostimulation in HD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002679
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Hemodialysis Complication
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diabetic HD group (Experimental): Patients of this group will receive 20 minutes of extra oral TENS over skin of bilateral parotid glands (3 sessions weekly for 3 weeks)
  Interventions: Device: TENS
- Nondiabetic goup (Active Comparator): Patients of this group will receive 20 minutes of extra oral TENS over skin of bilateral parotid glands (3 sessions weekly for 3 weeks)
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — Patients of this group will receive 20 minutes of extra oral TENS over skin of bilateral parotid glands (3 sessions weekly for 3 weeks)

SUMMARY:
Xerostomia is a subjective complaint of dry mouth, whereas hyposalivation is an objective decreased of salivary flow. Hyposalivation was reported in 28.8 % of haemodialysis (HD) patients (Bruzda-Zwiech, 2014).

DETAILED DESCRIPTION:
Stimulation of the salivary glands can be induced mechanically (for example, by chewing gum or acupressure) or through medications (such as pilocarpine, cevimeline, angiotensin-converting-enzyme inhibitors and angiotensin-receptor blockers) or by electrostimulation as transcutnaeous electrical nerve stimulation (TENS) (Bossola and Tazza, 2012).

Eighty HD patients (40 diabetics and 40 nondiabetics) will receive 20 minutes of TENS on skin over bilateral parotid gland, 3 times weekly for 3 weeks to investigate the hyposalivation response of diabetic and non diabetic HD patients to TENS.

ELIGIBILITY:
Inclusion Criteria:

* Eighty HD patients (40 diabetics and 40 non diabetics)
* HD at least from three month
* saliva flow less than or equal 0.15 millilitre per minute

Exclusion Criteria:

* pulmonary or cardiac disorders
* drugs to treat hyposalivation
* salivary glands inflammation, tumor, and autoimmune diseases.
* smokers and alcholics

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 80 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
3-week response of salivary flow rate | immediately after the last session
  the patients will be ordered to spit saliva in a graduated test tube for 5 minutes after the last session (session number 9). To calculate salivary flow rate: saliva volume will be divided on duration of saliva spitting.

SECONDARY OUTCOMES:
immediate response of saliva flow | immediately after the first session
  the patients will be ordered to spit saliva in a graduated test tube for 5 minutes immediately after the first session . To calculate salivary flow rate: saliva volume will be divided on duration of saliva spitting.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Faculty of Physical Therapy Cairo University, Giza, Dokki
  - Cairo Unoversity, Giza